CLINICAL TRIAL: NCT06097624
Title: Effectiveness of Synchronized Tele-exercise on Sleep Quality and Quality of Life for Healthy Young Adults: A Randomized Double-blind Controlled Trial
Brief Title: Effectiveness of Synchronized Tele-exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Collaborators: Ankara Medipol University (Other); Istanbul University - Cerrahpasa (Other); Duha Saydam Physical Therapy and Clinical Pilates Center (name of the center) (Unknown); Ozel Uç Ufuk Çizgisi Special Education and Rehabilitation Center (name of the center (Unknown)
Responsible Party: Principal Investigator, Begüm Okudan, Researcher, Okan University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 223091
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Examiners and researchers who are going to run the data analysis will be blinded to the assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): The exercises will be applied three times a week for four weeks. Each exercise is going to start with 10 repetitions and 1 set in the first session, and the exercises will be revised at the beginning of each week. Resistance will gradually be increased, and after four weeks, 3 sets of 10 repetitions will be targeted.
  Interventions: Other: synchronized tele-exercise
- Control (No Intervention): After a waiting period of four weeks, the participants will be contacted for reevaluation, and at the end of the assessment, an individual home exercise program will be created for them.

INTERVENTIONS:
Other: synchronized tele-exercise — All evaluations and exercise interventions will be performed by via Google Meet, a video-conferencing application. The participation link will be sent to the individual by the researcher before each session. In case of any technological disruption, the session will be postponed to the nearest available time by phone. All interventions will be run by a blinded researcher.
  Arms: Exercise

SUMMARY:
The aim of this study is to determine the effect of telehealth-synchronized group exercise on sleep and quality of life, and secondarily, on the health and body perception of healthy young adults. This study is planned as a randomized double-blind controlled clinical study.

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of telehealth-synchronized group exercise on sleep and quality of life, and secondarily, on the health and body perception of healthy young adults. This study is planned as a randomized double-blind controlled clinical study. The sample size was calculated using G*power 3.1.9.2, which required 42 patients and a size effect of 0.8, 80% power, 1:1 allocation ratio, and an error probability of 0.05. Forty-eight participants were planned to be included in the study, based on the probability that 15% of the patients could be excluded.

ELIGIBILITY:
Inclusion Criteria:

* being a volunteer,
* being in the age range of 18-25,
* having no barriers to online sessions through a computer,
* having no visual impairment.

Exclusion Criteria:

* having experienced a physical injury in the last 3 months
* having any major disorder,
* learning difficulty,
* having a mental disorder that could affect the results

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | 0th week
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item self-report questionnaire that assesses sleep quality over the last month. Its adaptation to Turkish and its reliability and validity analyses were carried out in 1996 by Ağargün el al. It covers seven components of sleep each of which are scored between 0-3: sleep duration, sleep disturbances, sleep latency, daytime dysfunction due to sleepiness, sleep efficiency, overall sleep quality, and sleep medication use. The PSQI provides a global score that ranges from 0 to 21, with higher scores indicating poorer sleep quality: smaller than 5, the score points to "Good Sleep Quality"; greater than or equal to 5, it indicates poor sleep quality (Buysee 1989, Agargun 1996). PSQI is a reliable and valid tool for assessing sleep quality in clinical and research settings.
The Pittsburgh Sleep Quality Index (PSQI) | 4th week
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item self-report questionnaire that assesses sleep quality over the last month. Its adaptation to Turkish and its reliability and validity analyses were carried out in 1996 by Ağargün el al. It covers seven components of sleep each of which are scored between 0-3: sleep duration, sleep disturbances, sleep latency, daytime dysfunction due to sleepiness, sleep efficiency, overall sleep quality, and sleep medication use. The PSQI provides a global score that ranges from 0 to 21, with higher scores indicating poorer sleep quality: smaller than 5, the score points to "Good Sleep Quality"; greater than or equal to 5, it indicates poor sleep quality (Buysee 1989, Agargun 1996). PSQI is a reliable and valid tool for assessing sleep quality in clinical and research settings.
World Health Organization Quality of Life-Brief Form | 0th week
  The WHOQOL is based on a purely subjective evaluation to assess the perceived quality of life. The short version, the World Health Organization Quality of Life-Brief Form (WHOQOL-BREF) is a 26-item self-report questionnaire that assesses the quality of life (QOL) within the context of an individual's culture, value systems, personal goals, standards, and concerns. It covers four domains: physical health, psychological health, social relationships, and environmental health.
World Health Organization Quality of Life-Brief Form | 4th week
  The WHOQOL is based on a purely subjective evaluation to assess the perceived quality of life. The short version, the World Health Organization Quality of Life-Brief Form (WHOQOL-BREF) is a 26-item self-report questionnaire that assesses the quality of life (QOL) within the context of an individual's culture, value systems, personal goals, standards, and concerns. It covers four domains: physical health, psychological health, social relationships, and environmental health.

SECONDARY OUTCOMES:
Body Perception | 0th week
  Participants will be asked to choose how they perceived their current body image, or "how they look'. Body mass index (BMI) classification will be used: 'Underweight', 'Healthy weight', 'Overweight', 'Obese', 'Severely obese'.
Body Perception | 4th week
  Participants will be asked to choose how they perceived their current body image, or "how they look'. Body mass index (BMI) classification will be used: 'Underweight', 'Healthy weight', 'Overweight', 'Obese', 'Severely obese'.
Perception of General Health | 0th week
  Participants will be asked to rate their perceived general health using a 10-point Likert scale; 1 indicating 'Very poor', 10 indicating 'Excellent'.
Perception of General Health | 4th week
  Participants will be asked to rate their perceived general health using a 10-point Likert scale; 1 indicating 'Very poor', 10 indicating 'Excellent'.
Perception of Physical Fitness | 0th week
  Participants will be asked to rate their perceived physical fitness using a 10-point Likert scale; 1 indicating 'Very poor', 10 indicating 'Excellent'.
Perception of Physical Fitness | 4th week
  Participants will be asked to rate their perceived physical fitness using a 10-point Likert scale; 1 indicating 'Very poor', 10 indicating 'Excellent'.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Okan University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No